CLINICAL TRIAL: NCT04032704
Title: Open-Label Phase 2 Study of Ladiratuzumab Vedotin (LV) for Unresectable Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of Ladiratuzumab Vedotin in Advanced Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed due to portfolio prioritization
Sponsor: Seagen Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGNLVA-005
Expanded Access: NCT06362590 (Available)
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Small Cell Lung Cancer; Non-small Cell Lung Cancer, Squamous; Non-small Cell Lung Cancer, Non-squamous; Head and Neck Squamous Cell Carcinoma; Esophageal Squamous Cell Carcinoma; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Prostate Cancer; Melanoma
Keywords: SCLC; NSCLC-squamous; NSCLC-nonsquamous; HNSCC; GEJ adenocarcinoma; Seattle Genetics
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma; Prostatic Neoplasms; Melanoma | interventions — SGN-LIV1A; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Non-randomized LV monotherapy (Experimental): Monotherapy dosing schedule 1.
  Interventions: Drug: ladiratuzumab vedotin
- Part B: Non-randomized LV monotherapy (Experimental): Monotherapy dosing schedule 2.
  Interventions: Drug: ladiratuzumab vedotin
- Part C - Arm 1: Randomized LV monotherapy (Experimental): Monotherapy dosing schedule 3.
  Interventions: Drug: ladiratuzumab vedotin
- Part C - Arm 2: Randomized LV combination therapy (Experimental): Combination dosing schedule 1.
  Interventions: Drug: ladiratuzumab vedotin; Drug: pembrolizumab
- Part C - Arm 3: Randomized LV combination therapy (Experimental): Combination dosing schedule 2.
  Interventions: Drug: ladiratuzumab vedotin; Drug: pembrolizumab

INTERVENTIONS:
Drug: ladiratuzumab vedotin — Intravenous (into the vein; IV) infusion
  Other Names: SGN-LIV1A
Drug: pembrolizumab — 200mg given by IV on Day 1 of each 21-day cycle
  Other Names: Keytruda
  Arms: Part C - Arm 2: Randomized LV combination therapy; Part C - Arm 3: Randomized LV combination therapy

SUMMARY:
This trial will study ladiratuzumab vedotin (LV) alone and with pembrolizumab to find out if it works to treat different types of solid tumors. It will also find out what side effects may occur. A side effect is anything the drug does besides treating cancer.

DETAILED DESCRIPTION:
This trial is designed to assess the antitumor activity, safety, and tolerability of LV alone and with pembrolizumab, for the treatment of solid tumors. Participants with the following advanced solid tumors will be enrolled:

Cohort 1: small cell lung cancer (SCLC) Cohort 2: non-small cell lung cancer-squamous (NSCLC-squamous) Cohort 3: non-small cell lung cancer-nonsquamous (NSCLC-nonsquamous) Cohort 4: head and neck squamous cell carcinoma (HNSCC) Cohort 5: esophageal squamous cell carcinoma (esophageal-squamous) Cohort 6: gastric and gastroesophageal junction (GEJ) adenocarcinoma Cohort 7: castration-resistant prostate cancer (CRPC) Cohort 8: melanoma

Participants will continue to receive study treatment until disease progression, unacceptable toxicity, investigator decision, consent withdrawal, study termination by the sponsor, pregnancy, or death, whichever comes first.

ELIGIBILITY:
Inclusion Criteria

* All Cohorts

  * Measurable disease according to RECIST v1.1 as assessed by the investigator
  * Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1
* Cohort 1: SCLC (Parts A and B)

  * Must have extensive stage disease
  * Must have disease progression during or following prior platinum-based systemic chemotherapy for extensive stage disease;
  * No more than 1 prior line of cytotoxic chemotherapy for extensive disease stage
  * May have received prior anti-PD(L)1 therapy
* Cohort 2: NSCLC-squamous (Parts A and B)

  * Must have unresectable locally advanced or metastatic disease
  * Must have disease progression during or following systemic therapy

    * Participants must have progressed during or after a platinum-based combination therapy administered for the treatment of metastatic disease, OR
    * Participants must have progressed within 6 months of last dose of platinum-based adjuvant, neoadjuvant, or definitive chemotherapy, or concomitant chemoradiation regimen for early stage or locally advanced stage disease.
  * Participants with known epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), reactive oxygen species (ROS), BRAF, or other actionable mutations are not eligible
  * No more than 1 prior line of cytotoxic chemotherapy for their advanced disease
  * Must have received prior anti-PD(L)1 therapy, unless contraindicated
* Cohort 3: NSCLC-nonsquamous (Parts A and B)

  * Must have unresectable locally advanced or metastatic disease
  * Must have disease progression during or following systemic therapy

    * Participants must have progressed during or after a platinum-based combination therapy administered for the treatment of metastatic disease, OR
    * Participants must have progressed within 6 months of last dose of platinum-based adjuvant, neoadjuvant, or definitive chemotherapy, or concomitant chemoradiation regimen for early stage or locally advanced state disease.
  * Participants with known EGFR, ALK, ROS, BRAF, tropomyosin receptor kinase (TRK), or other actionable mutations are not eligible
  * Must have had prior platinum-based chemotherapy
  * No more than 1 prior line of cytotoxic chemotherapy for their advanced disease
  * Must have received prior anti-PD(L)1 therapy, unless contraindicated
* Cohort 4: HNSCC (Parts A and B)

  * Must have unresectable locally recurrent or metastatic disease

    * Must have disease progression during or following prior line of systemic therapy
    * Disease progression after treatment with a platinum-containing regimen for recurrent/metastatic disease; OR
    * Recurrence/progression within 6 months of last dose of platinum therapy given as part of a multimodal therapy in the curative setting
  * No more than 1 line of cytotoxic chemotherapy for their advanced disease
  * May have received prior anti-PD(L)1 therapy, unless contraindicated
* Cohort 5: esophageal-squamous (Parts A and B)

  * Must have unresectable locally advanced or metastatic disease
  * Must have disease progression during or following systemic therapy
  * Must have had prior platinum-based chemotherapy
  * No more than 1 line of cytotoxic chemotherapy for their advanced disease
* Cohort 6: gastric and GEJ adenocarcinoma (Parts A and B)

  * Must have unresectable locally advanced or metastatic disease
  * Must have received prior platinum-based therapy
  * Must have disease progression during or following systemic therapy
  * Participants with known human epidermal growth factor receptor 2 (HER2) overexpression must have received prior HER2-targeted therapy
  * No more than 1 line of prior cytotoxic chemotherapy for their advanced disease
  * Participants may have received prior anti-PD(L)1 therapy, unless contraindicated
* Cohort 7: CRPC (Part B only)

  * Must have histologically or cytologically confirmed adenocarcinoma of the prostate

    * Participants with components of small cell of neuroendocrine histology are excluded
  * Must have metastatic castration-resistant disease
  * Must have been ≥28 days between cessation of androgen receptor-targeted therapy and start of study treatment
  * Must have received no more than 1 prior line of androgen receptor-targeted therapy for metastatic castration-sensitive prostate cancer or CRPC
  * No prior cytotoxic chemotherapy in the metastatic CRPC setting

    * For participants who received cytotoxic chemotherapy in CSPC, at least 6 months must have elapsed between last dose of chemotherapy and start of study treatment
    * No more than 1 prior line of cytotoxic chemotherapy for CSPC
  * Participants with measurable disease are eligible if the following criteria are met:

    * A minimum starting PSA level ≥1.0 ng/mL
    * Participants with measurable soft tissue disease must have evidence of measurable soft tissue disease according to PCWG3 criteria.
  * Participants with known breast cancer gene (BRCA) mutations are excluded
  * No prior radioisotope therapy or radiotherapy to ≥30% of bone marrow
* Cohort 8: Melanoma (Parts B and C)

  * Must have histologically or cytologically confirmed cutaneous malignant melanoma

    * Participants with mucosal, acral, or uveal melanoma are excluded
  * Must have locally advanced unresectable or metastatic stage disease
  * Must have progressive disease following anti-PD(L)1 therapy
  * Must have received BRAF +/- MEK inhibitor therapy if BRAF mutated (Part C)

Exclusion Criteria

* Active concurrent malignancy or a previous malignancy within the past 3 years
* Any anticancer therapy within 3 weeks of starting study treatment. Participants who are/were on adjuvant hormonal therapy for the treatment of malignancies with negligible risk of metastases are eligible.
* Known active central nervous system lesions
* Any ongoing clinically significant toxicity associated with prior treatment (Grade 2 or higher)
* Ongoing sensory or motor neuropathy of Grade ≥2
* Has received prior radiotherapy within 2 weeks of start of study treatment
* History of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (66):
- United States (27):
  - Ironwood Cancer & Research Centers - Chandler, Chandler, Arizona
  - Adventist Health White Memorial, Los Angeles, California
  - Providence Medical Foundation, Santa Rosa, California
  - Eastern CT Hematology and Oncology Associates, Norwich, Connecticut
  - GenesisCare USA, Jacksonville, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - IACT Health, Columbus, Georgia
  - Northwestern University, Chicago, Illinois
  - Decatur Memorial Hospital - Illinois, Decatur, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - University of Maryland, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - HealthPartners Institute, Saint Louis Park, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Valley Hospital, The / Luckow Pavilion, Paramus, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Weill Cornell Medicine, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - FirstHealth of the Carolinas, Pinehurst, North Carolina
  - Gabrail Cancer Center Research, LLC, Canton, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Saint Francis Hospital / Bon Secours - South Carolina, Greenville, South Carolina
  - Erlanger Oncology and Hematology, Chattanooga, Tennessee
  - Tennessee Oncology-Nashville/Sarah Cannon Research Institute, Nashville, Tennessee
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - UT Health East Texas Hope Cancer Center, Tyler, Texas
  - Carbone Cancer Center / University of Wisconsin, Madison, Wisconsin
- Australia (8):
  - Flinders Medical Centre, Bedford Park, Other
  - Townsville Cancer Center, Douglas, Other
  - Peninsula and South East Oncology, Frankston, Other
  - Central Coast Local Health District (Gosford and Wyong Hospitals), Gosford, Other
  - Royal Hobart Hospital, Hobart, Other
  - Cabrini, Malvern, Other
  - St Vincents Hospital Sydney, Sydney, Other
  - Melanoma Institute Australia, Wollstonecraft, Other
- Italy (11):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna, Other
  - Azienda Ospedaliero Universitaria Careggi, Florence, Other
  - ASL 3 Genovese Villa Scassi Hospital, Genova, Other
  - San Luca Hospital, Lucca, Other
  - Irccs Irst, Meldola, Other
  - Niguarda Ca' Granda Hospital, Milan, Other
  - Istituto Europeo di Oncologia, Milan, Other
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Other
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli, Other
  - Policlinico Universitario Agostino Gemelli, Roma, Other
  - AOUS Policlinico Le Scotte, Siena, Other
- South Korea (10):
  - Dong-A University Hospital, Busan, Other
  - Chonnam National University Hwasun Hospital, Hwasun, Other
  - Seoul National University Bundang Hospital, Seongnam-si, Other
  - Seoul National University Hospital, Seoul, Other
  - Severance Hospital, Yonsei University Health System, Seoul, Other
  - Samsung Medical Center, Seoul, Other
  - Seoul National University Boramae Medical Center, Seoul, Other
  - Korea University Guro Hospital, Seoul, Other
  - St. Vincent's Hospital, The Catholic University of Korea, Suwon, Other
  - Ajou University Hospital, Suwon, Other
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung, Other
  - National Cheng-Kung University Hospital, Tainan, Other
  - National Taiwan University Hospital, Taipei, Other
  - Taipei Medical University Hospital, Taipei, Other
- United Kingdom (6):
  - The Beatson West of Scotland Cancer Centre, Glasgow, Other
  - The Royal Marsden Hospital, London, Other
  - Sarah Cannon Research Institute UK, London, Other
  - UCL Cancer Institute, London, Other
  - The Christie NHS Foundation Trust, Manchester, Other
  - The Royal Marsden Hospital (Surrey), Sutton, Other

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had Parts A, B and C. Study was terminated and Part C was not opened. A total of 205 participants were enrolled in Part A (49 participants) and Part B (156 participants) of this study. In Part A all enrolled participants received study intervention while in Part B, 2 participants did not receive study intervention.
Pre-assignment Details: Cohorts of study: Cohort 1: small cell lung cancer (SCLC) (Part A, B); Cohort 2: non-SCLC-squamous (NSCLC-squamous) (Part A, B); Cohort 3: NSCLC-nonsquamous (Part A, B); Cohort 4: head & neck squamous cell carcinoma (HNSCC) (Part A, B); Cohort 5: esophageal squamous cell carcinoma (esophageal-squamous) (Part A, B); Cohort 6: gastric & gastroesophageal junction (GEJ) adenocarcinoma (Part A, B); Cohort 7: castration-resistant prostate cancer (CRPC) (Part B); Cohort 8: melanoma (Part B).
Groups:
- Part A: Cohort 1, LV 2.5 mg/kg: Participants with SCLC were administered ladiratuzumab vedotin (LV) 2.5 milligram per kilogram (mg/kg) as intravenous (IV) fusion on Day 1 of each 21-day cycle (q3wk) .
- Part A: Cohort 2, LV 2.5 mg/kg: Participants with NSCLC-squamous were administered LV 2.5 mg/kg as IV fusion q3wk.
- Part A: Cohort 3, LV 2.5 mg/kg: Participants with NSCLC-nonsquamous were administered LV 2.5 mg/kg as IV fusion q3wk.
- Part A: Cohort 4, LV 2.5 mg/kg: Participants with HNSCC were administered LV 2.5 mg/kg as IV fusion q3wk.
- Part A: Cohort 5, LV 2.5 mg/kg: Participants with esophageal-squamous were administered LV 2.5 mg/kg as IV fusion q3wk.
- Part A: Cohort 6, LV 2.5 mg/kg: Participants with GEJ were administered LV 2.5 mg/kg as IV fusion q3wk.
- Part B: Cohort 1, LV 1.25 mg/kg: Participants with SCLC were administered LV 1.25 mg/kg on Days 1, 8 and 15 of each 21-day cycle (q1wk) as a 30-minute IV infusion.
- Part B: Cohort 2, LV 1.25 mg/kg: Participants with NSCLC-squamous were administered LV 1.25 mg/kg on Days 1, 8 and 15 q1wk as a 30-minute IV infusion.
- Part B: Cohort 3, LV 1.25 mg/kg: Participants with NSCLC-nonsquamous were administered LV 1.25 mg/kg on Days 1, 8 and 15 q1wk as a 30-minute IV infusion.
- Part B: Cohort 4, LV 1.25 mg/kg: Participants with HNSCC were administered LV 1.25 mg/kg on Days 1, 8 and 15 q1wk as a 30-minute IV infusion.
- Part B: Cohort 5, LV 1.25 mg/kg: Participants with esophageal-squamous were administered LV 1.25 mg/kg on Days 1, 8 and 15 q1wk as a 30-minute IV infusion.
- Part B: Cohort 6, LV 1.25 mg/kg: Participants with GEJ were administered LV 1.25 mg/kg on Days 1, 8 and 15 q1wk as a 30-minute IV infusion.
- Part B: Cohort 7, LV 1.25 mg/kg: Participants with CRPC were administered LV 1.25 mg/kg on Days 1, 8 and 15 q1wk as a 30-minute IV infusion.
- Part B: Cohort 8, LV 1.25 mg/kg: Participants with melanoma were administered LV 1.25 mg/kg on Days 1, 8 and 15 q1wk as a 30-minute IV infusion.
- Part B: Cohort 1, LV 1.0 mg/kg: Participants with SCLC were administered LV 1.0 mg/kg q1wk on Days 1, 8 and 15 as a 30-minute IV infusion.
- Part B: Cohort 3, LV 1.0 mg/kg: Participants with NSCLC-nonsquamous were administered LV 1.0 mg/kg on Days 1, 8 and 15 q1wk as a 30-minute IV infusion.
- Part B: Cohort 4, LV 1.0 mg/kg: Participants with HNSCC were administered LV 1.0 mg/kg on Days 1, 8 and 15 q1wk as a 30-minute IV infusion.
- Part B: Cohort 6, LV 1.0 mg/kg: Participants with GEJ were administered LV 1.0 mg/kg on Days 1, 8 and 15 q1wk as a 30-minute IV infusion.
Period: Part A
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Started | 10 | 2 | 13 | 7 | 5 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 2 | 13 | 7 | 5 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0 | 1 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 9 | 2 | 10 | 7 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 16 (Participants were enrolled in Part-B of the study.) | 16 (Participants were enrolled in Part-B of the study.) | 19 (Participants were enrolled in Part-B of the study.) | 14 (Participants were enrolled in Part-B of the study.) | 17 (Participants were enrolled in Part-B of the study.) | 21 (Participants were enrolled in Part-B of the study.) | 14 (Participants were enrolled in Part-B of the study.) | 31 (Participants were enrolled in Part-B of the study.) | 2 (Participants were enrolled in Part-B of the study.) | 2 (Participants were enrolled in Part-B of the study.) | 2 (Participants were enrolled in Part-B of the study.) | 2 (Participants were enrolled in Part-B of the study.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 16 | 19 | 14 | 17 | 21 | 14 | 31 | 2 | 2 | 2 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 5 | 13 | 0 | 0 | 0 | 0
Not completed — Study termination by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 1 | 4 | 6 | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 13 | 14 | 12 | 12 | 13 | 7 | 17 | 2 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received any amount of study drug.
Groups:
- Part A: Cohort 1, LV 2.5 mg/kg: Participants with SCLC were administered ladiratuzumab vedotin (LV) 2.5 milligram per kilogram (mg/kg) as intravenous (IV) fusion on Day 1 of each 21-day cycle (q3wk).
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg | Total
Number analyzed (Participants) | 10 | 2 | 13 | 7 | 5 | 12 | 16 | 16 | 19 | 14 | 17 | 21 | 13 | 30 | 2 | 2 | 2 | 2 | 203
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (9.5) | 80.5 (4.9) | 67.2 (13.7) | 63.1 (12.3) | 70.8 (11.2) | 64.7 (10.3) | 65.0 (10.7) | 67.3 (8.8) | 63.9 (9.3) | 63.8 (9.9) | 60.5 (8.3) | 60.9 (8.9) | 71.9 (8.5) | 63.4 (12.2) | 61.0 (1.4) | 66.0 (2.8) | 56.0 (2.8) | 77.5 (6.4) | 64.7 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 8 | 2 | 1 | 0 | 7 | 4 | 5 | 3 | 2 | 3 | 0 | 7 | 0 | 1 | 0 | 0 | 46
  Male | 8 | 1 | 5 | 5 | 4 | 12 | 9 | 12 | 14 | 11 | 15 | 18 | 13 | 23 | 2 | 1 | 2 | 2 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 10 | 2 | 13 | 7 | 5 | 12 | 15 | 13 | 18 | 14 | 14 | 16 | 12 | 27 | 2 | 1 | 2 | 2 | 185
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 3 | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 2 | 1 | 4 | 8 | 2 | 1 | 3 | 1 | 9 | 4 | 0 | 3 | 0 | 0 | 0 | 0 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5
  White | 5 | 2 | 10 | 6 | 1 | 4 | 14 | 13 | 14 | 11 | 5 | 12 | 10 | 25 | 2 | 2 | 2 | 2 | 140
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 5 | 2 | 2 | 0 | 0 | 0 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Part A: Confirmed Objective Response Rate (ORR) as Determined by Investigator According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Confirmed ORR was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) per RECIST v.1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to less than (<) 10 millimeter (mm). PR was defined as more than or equal to (>=) 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Participants who did not have at least 2 post-baseline response assessment (initial response and confirmation scan) were counted as non-responders.
Time Frame: From the first dose of study treatment until the first documented CR or PR or new anticancer therapies or death, whichever occurred first (maximum up to 8.3 months)
Population: The full analysis set (FAS) included all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 10 | 2 | 13 | 7 | 5 | 12
Percentage of participants | 10 [0.3 to 44.5] | 0 [0.0 to 84.2] | 8 [0.2 to 36.0] | 14 [0.4 to 57.9] | 20 [0.5 to 71.6] | 8 [0.2 to 38.5]

2. Primary Outcome: Part B: Confirmed ORR as Determined by Investigator According to RECIST v1.1
Description: Confirmed ORR was defined as the percentage of participants with a confirmed CR or PR per RECIST v.1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm. PR was defined as >= 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Participants who did not have at least 2 post-baseline response assessment (initial response and confirmation scan) were counted as non-responders.
Time Frame: From the first dose of study treatment until the first documented CR or PR or new anticancer therapies or death, whichever occurred first (maximum up to 34.7 months for 1.25 mg/kg and 5.7 months for 1 mg/kg dose level)
Population: The FAS included all participants who received any amount of study drug. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 16 | 16 | 19 | 14 | 17 | 21 | 13 | 30 | 2 | 2 | 2 | 2
Percentage of participants | 6 [0.2 to 30.2] | 13 [1.6 to 38.3] | 11 [1.3 to 33.1] | 0 [0.0 to 23.2] | 18 [3.8 to 43.4] | 14 [3.0 to 36.3] | 0 [0.0 to 24.7] | 20 [7.7 to 38.6] | 0 [0.0 to 84.2] | 0 [0.0 to 84.2] | 0 [0.0 to 84.2] | 50 [1.3 to 98.7]

3. Primary Outcome: Part B: Confirmed Prostate-Specific Antigen (PSA) Response Rate as Determined by Investigator According to Prostate Cancer Clinical Trials Working Group 3 (PCWG3) Criteria, for Prostate Cancer
Description: Confirmed PSA response rate was defined as the percentage of participants with a reduction from baseline PSA level of at least 50%, measured twice >= 3 weeks apart. PSA progression was defined as per PCWG3 criteria- a) if a participant presented first a decline from baseline, progression was defined as the first PSA increase that was >=25% and >=2 nanograms per milliliter (ng/mL) above the nadir, and which was confirmed by a consecutive second value >=3 weeks later that fulfilled the same criteria (that is, a confirmed rising trend); b) if a participant did not present a decline from baseline, progression was defined as the first PSA increase that was >=25% and >=2 ng/mL increased from baseline beyond 12 weeks.
Time Frame: From the first dose of study treatment up to the date of last response assessment (maximum up to 13.5 months)
Population: The FAS included all participants who received any amount of study drug. As prespecified in protocol, this outcome measure was planned to be analyzed only in the Part B: Cohort 7, LV 1.25 mg/kg arm. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Cohort 7, LV 1.25 mg/kg
Number analyzed (Participants) | 13
Percentage of participants | 23 [5.0 to 53.8]

4. Secondary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs), Treatment Related TEAEs and >= Grade 3 TEAE
Description: An adverse event (AE) was any untoward medical occurrence in a participant/ clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. AEs included both SAEs ad all non-SAEs. TEAEs were defined as newly occurring (not present at baseline)/worsening after first dose of study treatment. TESAEs were any untoward medical occurrence at any dose that: suspected to cause death; life-threatening; required hospitalization; persistent/significant disability/incapacity & may cause congenital anomaly/birth defect. Treatment related TEAEs were related to study treatment and relatedness was judged by investigator. TEAEs were graded according to National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version (v) 4.03 (grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening).
Time Frame: From start of study treatment up to 30 days after last dose of study treatment (maximum up to 37.5 months)
Population: The safety analysis set included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 10 | 2 | 13 | 7 | 5 | 12
Participants
  TEAEs | 10 | 2 | 13 | 7 | 5 | 12
  TESAEs | 5 | 1 | 7 | 2 | 3 | 3
  Treatment Related TEAEs | 9 | 2 | 11 | 7 | 5 | 11
  TEAEs (>= Grade 3) | 7 | 1 | 9 | 4 | 4 | 6

5. Secondary Outcome: Part B: Number of Participants With TEAEs, TESAEs, Treatment Related TEAEs and >= Grade 3 TEAE
Description: An AE was any untoward medical occurrence in a participant, or a clinical investigational participant administered a medicinal product, and which does not necessarily have a causal relationship with this treatment. AEs included both SAEs ad all non-SAEs. TEAEs were defined as newly occurring (not present at baseline) or worsening after first dose of study treatment. TESAEs were any untoward medical occurrence at any dose that: suspected to cause death; life-threatening; required hospitalization; persistent or significant disability or incapacity and may cause congenital anomaly or birth defect. Treatment related TEAEs were related to study treatment and relatedness was judged by investigator. TEAEs were graded according to NCI-CTCAE v4.03 (grade 1= mild, grade 2= moderate, grade 3= severe and grade 4= life-threatening).
Time Frame: From start of study treatment up to 30 days after last dose of study treatment (maximum up to 37.5 months)
Population: The safety analysis set included all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 16 | 16 | 19 | 14 | 17 | 21 | 13 | 30 | 2 | 2 | 2 | 2
Participants
  TEAEs | 15 | 16 | 19 | 14 | 17 | 21 | 13 | 30 | 2 | 2 | 2 | 2
  TESAEs | 6 | 5 | 9 | 8 | 9 | 12 | 4 | 11 | 1 | 2 | 1 | 0
  Treatment Related TEAEs | 13 | 16 | 18 | 12 | 17 | 19 | 12 | 28 | 2 | 2 | 2 | 2
  TEAEs (>= Grade 3) | 12 | 11 | 14 | 11 | 13 | 17 | 8 | 17 | 1 | 2 | 1 | 0

6. Secondary Outcome: Part A: Confirmed Investigator Determined Disease Control Rate (DCR) According to RECIST v1.1
Description: DCR was defined as percentage of participants who achieved confirmed and unconfirmed CR or PR per RECIST v1.1 or met stable disease (SD) criteria at least once after start of study treatment at minimum interval of 5 weeks. CR was defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR was defined as >= 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference smallest sum diameters while on study. PD: at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study (this included baseline sum if that is smallest on study). In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 0.5 cm. Appearance of one or more new lesions was also considered progression.
Time Frame: From the first dose of study treatment until the first documented CR, PR or SD or new anticancer therapies or death, whichever occurred first (maximum up to 4.1 months)
Population: The FAS included all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 10 | 2 | 13 | 7 | 5 | 12
Percentage of participants | 40 [12.2 to 73.8] | 50 [1.3 to 98.7] | 46 [19.2 to 74.9] | 57 [18.4 to 90.1] | 60 [14.7 to 94.7] | 33 [9.9 to 65.1]

7. Secondary Outcome: Part B: Confirmed Investigator Determined DCR According to RECIST v1.1
Description: DCR was defined as percentage of participants who achieved confirmed and unconfirmed CR or PR per RECIST v1.1 or met SD criteria at least once after start of study treatment at a minimum interval of 5 weeks. CR was defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR was defined as >= 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: At least 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 0.5 centimeter (cm). Appearance of one or more new lesions was also considered progression.
Time Frame: From the first dose of study treatment until the first documented CR, PR or SD or new anticancer therapies or death, whichever occurred first (maximum up to 5.5 months for 1.25 mg/kg and 1.5 months for 1 mg/kg dose level)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 16 | 16 | 19 | 14 | 17 | 21 | 13 | 30 | 2 | 2 | 2 | 2
Percentage of participants | 19 [4.0 to 45.6] | 50 [24.7 to 75.3] | 58 [33.5 to 79.7] | 64 [35.1 to 87.2] | 59 [32.9 to 81.6] | 52 [29.8 to 74.3] | 62 [31.6 to 86.1] | 77 [57.7 to 90.1] | 50 [1.3 to 98.7] | 50 [1.3 to 98.7] | 0 [0.0 to 84.2] | 100 [15.8 to 100.0]

8. Secondary Outcome: Part A: Confirmed Investigator Determined Duration of Response (DOR) According to RECIST v1.1
Description: DOR:time from 1st documentation of OR(confirmed CR/PR per RECIST Version 1.1) to 1st documentation of PD/death due to any cause,whichever occurred first.CR:disappearance of all target lesions.Any pathological lymph nodes must have reduction in short axis to <10 mm.PR:>=30 % decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. Participants do not have PD and are still on study at time of analysis/are removed from study prior to documentation of PD were censored at last disease assessment documenting absence of PD. Participants who started new anticancer treatment prior to documentation of PD were censored at last disease assessment prior to start of new treatment.PD:at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study.In addition to relative increase of 20%, sum must demonstrate absolute increase of 0.5 cm.Appearance of one/more new lesions was considered progression. Kaplan-Meier method was used.
Time Frame: From the first documentation of CR or PR to PD or death or censoring whichever occurred first (maximum up to 5.7 months)
Population: The FAS included all participants who received any amount of study drug. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure. No participant had CR or PR in Part A: Cohort 2, LV 2.5 mg/kg arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1
Months | 5.7 [NA to NA] — There was only 1 participant evaluable, hence lower and upper limit of the 95% confidence interval could not be estimated. |  | 5.5 [NA to NA] — There was only 1 participant evaluable, hence lower and upper limit of the 95% confidence interval could not be estimated. | 3.7 [NA to NA] — There was only 1 participant evaluable, hence lower and upper limit of the 95% confidence interval could not be estimated. | 2.7 [NA to NA] — There was only 1 participant evaluable, hence lower and upper limit of the 95% confidence interval could not be estimated. | NA [NA to NA] — No participant had an event of interest; hence results could not be estimated.

9. Secondary Outcome: Part B: Confirmed Investigator Determined DOR According to RECIST v1.1
Description: as for outcome 8
Time Frame: From the first documentation of CR or PR to PD or death or censoring whichever occurred first (maximum up to 32.0 months for 1.25 mg/kg and 4.2 months for 1 mg/kg dose level)
Population: The FAS included all participants who received any amount of study drug. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure. No participant had CR or PR in Part B: Cohort 4, LV 1.25 mg/kg arm, Part B: Cohort 7, LV 1.25 mg/kg arm, Part B: Cohort 1, LV 1.0 mg/kg arm, Part B: Cohort 3, LV 1.0 mg/kg arm and Part B: Cohort 4, LV 1.0 mg/kg arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 1 | 2 | 2 | 0 | 3 | 3 | 0 | 6 | 0 | 0 | 0 | 1
Months | NA [NA to NA] — No participant had an event of interest; hence data could not be reported. | 7.5 [5.78 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. | NA [16.59 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. |  | NA [3.06 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. | 3.9 [2.60 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. |  | 8.3 [5.62 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. |  |  |  | 4.2 [NA to NA] — There was only 1 participant evaluable, hence lower and upper limit of the 95% confidence interval could not be estimated.

10. Secondary Outcome: Part B: Confirmed Investigator Determined PSA-DOR, for Prostate Cancer
Description: PSA-DOR was defined as the time from the first documentation of PSA response (subsequently confirmed at least 3 weeks apart) to the first documentation of PSA progression or death due to any cause, whichever occurred first. Confirmed PSA response rate was defined as the percentage of participants with a reduction from baseline PSA level of at least 50%, measured twice >= 3 weeks apart. Participants who do not have PD and are still on study at the time of an analysis or who are removed from the study prior to documentation of PD was censored at the date of last disease assessment documenting absence of PD. Participants who started a new anticancer treatment prior to documentation of PD were censored at the date of last disease assessment prior to the start of new treatment. The confidence interval (CI) was calculated using the complementary log-log transformation method.
Time Frame: From the first documentation of CR or PR to PD or death or censoring whichever occurred first (maximum up to 3 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Cohort 7, LV 1.25 mg/kg
Number analyzed (Participants) | 3
Months | 3.0 [1.9 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval.

11. Secondary Outcome: Part A: Confirmed Investigator Determined Progression Free Survival (PFS) According to RECIST v1.1
Description: PFS: time from start of study treatment to the first documentation of PD by RECIST v1.1 or clinical PD. Participants who do not have PD and are still on study at the time of an analysis or who are removed from the study prior to documentation of PD were censored at the date of last disease assessment documenting absence of PD. Participants who started a new anticancer treatment prior to documentation of PD were censored at the date of last disease assessment prior to the start of new treatment. PD: At least 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 0.5 cm. Appearance of one or more new lesions was also considered progression. Median was estimated using the Kaplan-Meier method and the CI was calculated using the complementary log-log transformation method.
Time Frame: From first dose of study treatment to the date of PD or clinical PD or censoring whichever occurred first (maximum up to 8.3 months)
Population: The FAS included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 10 | 2 | 13 | 7 | 5 | 12
Months | 1.4 [0.53 to 2.69] | 1.5 [1.25 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. | 2.5 [0.46 to 4.17] | 2.3 [0.33 to 4.86] | 2.9 [0.59 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. | 1.4 [1.31 to 4.17]

12. Secondary Outcome: Part B: Confirmed Investigator Determined PFS According to RECIST v1.1
Description: as for outcome 11
Time Frame: From first dose of study treatment to the date of PD or clinical PD or censoring whichever occurred first (maximum up to 34.7 months for 1.25 mg/kg and 5.7 months for 1 mg/kg dose level)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 16 | 16 | 19 | 14 | 17 | 21 | 13 | 30 | 2 | 2 | 2 | 2
Months | 1.4 [1.18 to 2.04] | 1.8 [1.12 to 5.72] | 2.4 [1.31 to 2.96] | 2.7 [1.18 to 2.86] | 2.8 [1.38 to 3.32] | 2.3 [1.25 to 2.73] | 4.9 [2.10 to 5.65] | 4.2 [2.50 to 6.97] | 1.9 [1.02 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. | NA [NA to NA] — Only one participant had event, hence median and CI were not reported. The individual participant data was 1.3 months. | 1.5 [1.35 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. | 4.2 [2.76 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval.

13. Secondary Outcome: Part B: Confirmed Investigator Determined PSA-PFS, for Prostate Cancer
Description: PSA-PFS: time from start of study treatment to first documentation of PSA progression or death due to any cause, whichever occurred first. Participants who do not have PD and are still on study at time of analysis or who are removed from study prior to documentation of PD was censored at date of last disease assessment documenting absence of PD. Participants who started new anticancer treatment prior to documentation of PD were censored at date of last disease assessment prior to the start of new treatment. PD: at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study (this included baseline sum if that is smallest on study). In addition to relative increase of 20%, sum must also demonstrate absolute increase of at least 0.5 cm. Appearance of one or more new lesions was also considered progression. Median was estimated using Kaplan-Meier method and CI was calculated using the complementary log-log transformation method.
Time Frame: From first dose of study treatment to the date of PD or clinical PD or censoring whichever occurred first (maximum up to 5.7 months)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Cohort 7, LV 1.25 mg/kg
Number analyzed (Participants) | 9
Months | 3.7 [2.8 to 5.1]

14. Secondary Outcome: Part A: Overall Survival (OS)
Description: OS was defined as the time from the start of study treatment to date of death due to any cause. Participants who do not have PD and are still on study at the time of an analysis or who are removed from the study prior to documentation of PD was censored at the date of last disease assessment documenting absence of PD. Participants who started a new anticancer treatment prior to documentation of PD were censored at the date of last disease assessment prior to the start of new treatment. Median was estimated using the Kaplan-Meier method.
Time Frame: From first dose of study treatment to the date of death or censoring whichever occurred first (maximum up to 27.5 months)
Population: The FAS included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 10 | 2 | 13 | 7 | 5 | 12
Months | 6.1 [1.38 to 15.84] | 2.5 [1.74 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. | 6.5 [2.20 to 16.95] | 4.8 [0.33 to 6.97] | 7.2 [0.59 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. | 8.7 [3.98 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval.

15. Secondary Outcome: Part B: Overall Survival
Description: as for outcome 14
Time Frame: From first dose of study treatment to the date of death or censoring whichever occurred first (maximum up to 37.5 months for 1.25 mg/kg and 20.9 months for 1 mg/kg dose level)
Population: The FAS included all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 16 | 16 | 19 | 14 | 17 | 21 | 13 | 30 | 2 | 2 | 2 | 2
Months | 4.7 [3.45 to 8.74] | 9.0 [4.53 to 12.68] | 9.3 [2.92 to 20.14] | 5.2 [3.42 to 18.33] | 12.7 [4.17 to 15.28] | 3.8 [1.77 to 8.61] | 10.1 [6.47 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. | 11.5 [9.26 to 15.41] | 11.1 [1.22 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. | NA [1.71 to NA] — Insufficient number of participants with events to calculate the median and upper limit of the 95% confidence interval. | 5.6 [1.64 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval. | 14.2 [8.34 to NA] — Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval.

16. Secondary Outcome: Part A: Area Under the Serum Concentration Time Curve Between Days 0 to 21 (AUC21) of Ladiratuzumab Vedotin
Description: Area under the observed concentration-time curve from the time of dosing to Day 21 of LV was calculated by noncompartmental analysis.
Time Frame: AUC21 is reported on Day 21 using PK concentrations assessed at Pre-dose, end of infusion, 2 hour, 4 hour, 48 hour, 168 hour and 336 hour post dose of Cycle 1 (each cycle = 21 days, LV administered on Day 1 of cycle)
Population: The safety analysis set included all participants who received any amount of study drug. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 10 | 2 | 11 | 6 | 5 | 12
Day*micrograms per milliliter | 142.5 (18.9) | 175.6 (16.5) | 145.3 (35.1) | 146.6 (28.3) | 123.2 (21.7) | 132.0 (26.0)

17. Secondary Outcome: Part A: Maximum Serum Concentration (Cmax) According to Antibody-Drug Conjugate (ADC) Pharmacokinetic Parameters
Description: Cmax according to ADC pharmacokinetic parameters was reported.
Time Frame: Cmax during Day 1 to 21 post LV administration on Day 1 was reported using PK concentration assessed at Pre-dose, end of infusion, 2 hour, 4 hour, 48 hour, 168 hour and 336 hour post-dose of LV administration on Day 1 (each cycle = 21 days)
Population: The safety analysis set included all participants who received any amount of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 10 | 2 | 13 | 7 | 5 | 12
Micrograms per milliliter | 50.4 (31.2) | 58.6 (1.0) | 55.8 (29.6) | 52.3 (23.6) | 39.6 (14.7) | 55.2 (64.9)

18. Secondary Outcome: Part A: AUC21 of Total Antibody (TAB)
Description: Area under the observed concentration-time curve from the time of dosing to Day 21 of TAB was calculated by noncompartmental analysis.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 10 | 2 | 10 | 6 | 5 | 10
Day*micrograms per milliliter | 302.4 (19.7) | 328.5 (17.8) | 280.3 (34.1) | 292.3 (28.2) | 219.8 (28.5) | 258.9 (31.6)

19. Secondary Outcome: Part A: Cmax According to TAB Pharmacokinetic Parameters
Description: Cmax according to TAB pharmacokinetic parameters was reported.
Time Frame: as for outcome 17
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 9 | 2 | 11 | 7 | 5 | 10
Micrograms per milliliter | 61.6 (23.7) | 66.1 (20.8) | 68.2 (30.5) | 61.4 (16.1) | 50.7 (38.3) | 57.2 (24.1)

20. Secondary Outcome: Part A: AUC21 of Monomethyl Auristatin E (MMAE)
Description: Area under the observed concentration-time curve from the time of dosing to Day 21 of MMAE was calculated by noncompartmental analysis.
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*nanogram per milliliter
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 2 | 1 | 7 | 3 | 2 | 7
Day*nanogram per milliliter | 34.1 (21.1) | 50.5 (NA) — Insufficient number of participants to calculate the geometric coefficient of variation. | 62.9 (79.3) | 66.2 (45.6) | 91.0 (19.3) | 35.2 (36.9)

21. Secondary Outcome: Part A: Cmax According to MMAE Pharmacokinetic Parameters
Description: Cmax according to MMAE pharmacokinetic parameters was reported.
Time Frame: as for outcome 17
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 2 | 1 | 7 | 2 | 2 | 6
Nanogram per milliliter | 2.8 (15.7) | 5.7 (NA) — Insufficient number of participants to calculate the geometric coefficient of variation. | 6.4 (83.1) | 6.3 (10.6) | 11.3 (12.6) | 3.6 (41.8)

22. Secondary Outcome: Part B: Area Under the Concentration Time Curve Between Day 0 to 7 (AUC7) of ADC
Description: Area under the observed concentration-time curve from the time of dosing to Day 7 of ADC was calculated by noncompartmental analysis.
Time Frame: AUC7 is reported at Day 7 using PK concentration assessed at Pre-dose, end of infusion, 2hr, 4hr, 48hr post-dose of LV administration on Day 1; pre-dose PK concentration on Day 8 in Cycle 1 (each cycle=21 days, LV administered on Day 1, 8 and 15 of cycle)
Population: The safety analysis set included all participants who received any amount of study drug. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure. There were insufficient samples to provide pharmacokinetic (PK) estimates for analytes in Part B: Cohort 6, LV 1.0 mg/kg arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 14 | 11 | 18 | 9 | 14 | 12 | 11 | 25 | 2 | 2 | 1 | 0
Day*micrograms per milliliter | 57.3 (23.2) | 51.7 (16.9) | 59.5 (29.7) | 60.6 (36.7) | 43.3 (12.6) | 50.7 (27.2) | 66.0 (42.8) | 46.8 (25.0) | 42.1 (0.5) | 52.0 (0.1) | 44.8 (NA) — Insufficient number of participants to calculate the geometric coefficient of variation. |

23. Secondary Outcome: Part B: Cmax According to ADC Pharmacokinetic Parameters
Description: Cmax according to ADC pharmacokinetic parameters was reported.
Time Frame: Cmax during Day 1 to 7 post LV administration on Day 1 was reported using PK concentration assessed at Pre-dose, end of infusion, 2 hr, 4 hr, 48 hr post-dose of LV administration on Day 1 (each cycle = 21 days, LV administered on Day 1, 8 and 15 of cycle)
Population: The safety analysis set included all participants who received any amount of study drug. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure. There were insufficient samples to provide PK estimates for analytes in Part B: Cohort 6, LV 1.0 mg/kg arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 16 | 14 | 19 | 14 | 17 | 18 | 12 | 27 | 2 | 2 | 2 | 0
Micrograms per milliliter | 35.3 (35.0) | 27.8 (19.7) | 30.9 (19.2) | 28.7 (28.6) | 25.0 (28.8) | 28.0 (17.2) | 30.5 (15.1) | 25.4 (21.9) | 29.5 (20.3) | 24.3 (10.2) | 24.1 (6.2) |

24. Secondary Outcome: Part B: AUC7 of TAB
Description: Area under the observed concentration-time curve from the time of dosing to Day 7of TAB was calculated by noncompartmental analysis.
Time Frame: as for outcome 22
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 14 | 11 | 18 | 9 | 14 | 12 | 11 | 25 | 2 | 2 | 1 | 0
Day*micrograms per milliliter | 101.1 (29.4) | 92.7 (18.7) | 106.9 (29.8) | 91.2 (30.9) | 73.9 (20.7) | 85.7 (26.0) | 106.5 (28.2) | 74.7 (26.3) | 76.6 (22.6) | 88.6 (11.1) | 71.4 (NA) — Insufficient number of participants to calculate the geometric coefficient of variation. |

25. Secondary Outcome: Part B: Cmax According to TAB Pharmacokinetic Parameters
Description: Cmax according to TAB pharmacokinetic parameters was reported.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 16 | 14 | 19 | 14 | 17 | 17 | 12 | 29 | 2 | 2 | 2 | 0
Micrograms per milliliter | 38.3 (17.9) | 31.6 (16.6) | 36.8 (21.8) | 32.1 (26.2) | 27.4 (28.9) | 31.3 (19.7) | 32.6 (25.9) | 32.5 (73.8) | 26.8 (15.6) | 30.6 (14.8) | 27.9 (2.0) |

26. Secondary Outcome: Part B: AUC7 OF MMAE
Description: Area under the observed concentration-time curve from the time of dosing to Day 7 of MMAE was calculated by noncompartmental analysis.
Time Frame: as for outcome 22
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*micrograms per milliliter
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 14 | 11 | 18 | 9 | 14 | 12 | 11 | 25 | 2 | 2 | 1 | 0
Day*micrograms per milliliter | 14.6 (63.1) | 16.5 (55.6) | 11.9 (51.5) | 15.6 (51.0) | 17.3 (67.6) | 13.7 (83.0) | 10.7 (57.3) | 13.8 (45.2) | 10.8 (64.1) | 12.4 (25.9) | 8.5 (NA) — Insufficient number of participants to calculate the geometric coefficient of variation. |

27. Secondary Outcome: Part B: Cmax According to MMAE Pharmacokinetic Parameters
Description: Cmax according to MMAE pharmacokinetic parameters was reported.
Time Frame: Cmax during Day 1 to 7 post LV administration on Day 1 was reported using PK concentration assessed at Pre-dose, end of infusion, 2 hr, 4 hr, 48 hr post-dose of LV administration on Day 1 (each cycle= 21 days, LV administered on Day 1, 8 and 15 of cycle)
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 10 | 4 | 8 | 8 | 15 | 11 | 8 | 16 | 1 | 0 | 1 | 0
Nanograms per milliliter | 2.8 (60.7) | 4.5 (50.4) | 2.6 (59.1) | 2.7 (39.9) | 3.3 (65.8) | 2.9 (114.9) | 1.7 (28.9) | 2.4 (52.7) | 1.4 (NA) — Insufficient number of participants to calculate the geometric coefficient of variation. |  | 1.7 (NA) — Insufficient number of participants to calculate the geometric coefficient of variation. |

28. Secondary Outcome: Part A: Number of Participants With Positive Post-Baseline Antitherapeutic Antibody (ATA) Incidence
Description: A positive baseline ATA result was considered positive post-baseline if the post-baseline ATA titer result was at least four times higher than the baseline result.
Time Frame: From first ATA draw to last ATA draw (maximum up to 8.8 months)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg
Number analyzed (Participants) | 9 | 2 | 12 | 6 | 4 | 12
Participants
  Baseline Negative and Negative post-baseline | 8 | 2 | 9 | 4 | 4 | 10
  Baseline Negative and Positive post-baseline | 1 | 0 | 1 | 1 | 0 | 1
  Baseline Positive and Negative post-baseline | 0 | 0 | 2 | 1 | 0 | 1
  Baseline Positive and Positive post-baseline | 0 | 0 | 0 | 0 | 0 | 0

29. Secondary Outcome: Part B: Number of Participants With Positive Post-Baseline ATA Incidence
Description: as for outcome 28
Time Frame: From first ATA draw to last ATA draw (maximum up to 22.1 months for 1.25 mg/kg and 5.1 months for 1 mg/kg)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
Number analyzed (Participants) | 12 | 13 | 19 | 12 | 14 | 12 | 10 | 29 | 2 | 2 | 1 | 2
Participants
  Baseline Negative and Negative post-baseline | 10 | 11 | 13 | 12 | 11 | 10 | 9 | 24 | 2 | 0 | 1 | 2
  Baseline Negative and Positive post-baseline | 1 | 1 | 4 | 0 | 2 | 1 | 1 | 4 | 0 | 2 | 0 | 0
  Baseline Positive and Negative post-baseline | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Baseline Positive and Positive post-baseline | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 30 days after last dose of study treatment (maximum up to 37.5 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. All-cause mortality included all enrolled participants. SAEs and non-SAEs were analyzed in the safety analysis set. The safety analysis set included all participants who received any amount of study drug.
Arm/Group | Part A: Cohort 1, LV 2.5 mg/kg | Part A: Cohort 2, LV 2.5 mg/kg | Part A: Cohort 3, LV 2.5 mg/kg | Part A: Cohort 4, LV 2.5 mg/kg | Part A: Cohort 5, LV 2.5 mg/kg | Part A: Cohort 6, LV 2.5 mg/kg | Part B: Cohort 1, LV 1.25 mg/kg | Part B: Cohort 2, LV 1.25 mg/kg | Part B: Cohort 3, LV 1.25 mg/kg | Part B: Cohort 4, LV 1.25 mg/kg | Part B: Cohort 5, LV 1.25 mg/kg | Part B: Cohort 6, LV 1.25 mg/kg | Part B: Cohort 7, LV 1.25 mg/kg | Part B: Cohort 8, LV 1.25 mg/kg | Part B: Cohort 1, LV 1.0 mg/kg | Part B: Cohort 3, LV 1.0 mg/kg | Part B: Cohort 4, LV 1.0 mg/kg | Part B: Cohort 6, LV 1.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 9/10 | 2/2 | 10/13 | 7/7 | 4/5 | 5/12 | 13/16 | 13/16 | 14/19 | 12/14 | 12/17 | 13/21 | 7/13 | 16/30 | 2/2 | 1/2 | 2/2 | 2/2
Serious Adverse Events (participants affected / at risk) | 5/10 | 1/2 | 7/13 | 2/7 | 3/5 | 3/12 | 6/16 | 5/16 | 9/19 | 8/14 | 9/17 | 12/21 | 4/13 | 11/30 | 1/2 | 2/2 | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 10/10 | 2/2 | 13/13 | 6/7 | 5/5 | 12/12 | 15/16 | 16/16 | 19/19 | 14/14 | 17/17 | 19/21 | 13/13 | 30/30 | 2/2 | 2/2 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1, LV 2.5 mg/kg (N=10) | Part A: Cohort 2, LV 2.5 mg/kg (N=2) | Part A: Cohort 3, LV 2.5 mg/kg (N=13) | Part A: Cohort 4, LV 2.5 mg/kg (N=7) | Part A: Cohort 5, LV 2.5 mg/kg (N=5) | Part A: Cohort 6, LV 2.5 mg/kg (N=12) | Part B: Cohort 1, LV 1.25 mg/kg (N=16) | Part B: Cohort 2, LV 1.25 mg/kg (N=16) | Part B: Cohort 3, LV 1.25 mg/kg (N=19) | Part B: Cohort 4, LV 1.25 mg/kg (N=14) | Part B: Cohort 5, LV 1.25 mg/kg (N=17) | Part B: Cohort 6, LV 1.25 mg/kg (N=21) | Part B: Cohort 7, LV 1.25 mg/kg (N=13) | Part B: Cohort 8, LV 1.25 mg/kg (N=30) | Part B: Cohort 1, LV 1.0 mg/kg (N=2) | Part B: Cohort 3, LV 1.0 mg/kg (N=2) | Part B: Cohort 4, LV 1.0 mg/kg (N=2) | Part B: Cohort 6, LV 1.0 mg/kg (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngocele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute motor-sensory axonal neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Cohort 1, LV 2.5 mg/kg (N=10) | Part A: Cohort 2, LV 2.5 mg/kg (N=2) | Part A: Cohort 3, LV 2.5 mg/kg (N=13) | Part A: Cohort 4, LV 2.5 mg/kg (N=7) | Part A: Cohort 5, LV 2.5 mg/kg (N=5) | Part A: Cohort 6, LV 2.5 mg/kg (N=12) | Part B: Cohort 1, LV 1.25 mg/kg (N=16) | Part B: Cohort 2, LV 1.25 mg/kg (N=16) | Part B: Cohort 3, LV 1.25 mg/kg (N=19) | Part B: Cohort 4, LV 1.25 mg/kg (N=14) | Part B: Cohort 5, LV 1.25 mg/kg (N=17) | Part B: Cohort 6, LV 1.25 mg/kg (N=21) | Part B: Cohort 7, LV 1.25 mg/kg (N=13) | Part B: Cohort 8, LV 1.25 mg/kg (N=30) | Part B: Cohort 1, LV 1.0 mg/kg (N=2) | Part B: Cohort 3, LV 1.0 mg/kg (N=2) | Part B: Cohort 4, LV 1.0 mg/kg (N=2) | Part B: Cohort 6, LV 1.0 mg/kg (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 2 (3) | 0 (0) | 2 (3) | 2 (2) | 2 (4) | 6 (8) | 1 (1) | 7 (8) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 3 (4) | 4 (6) | 3 (3) | 2 (5) | 3 (3) | 1 (3) | 6 (8) | 2 (3) | 5 (8) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Androgen deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperprolactinaemia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (5) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 4 (6) | 6 (7) | 2 (4) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 1 (2) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 4 (6) | 3 (4) | 6 (8) | 5 (6) | 4 (6) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (9) | 3 (3) | 2 (2) | 4 (4) | 6 (8) | 9 (17) | 6 (11) | 5 (5) | 5 (7) | 8 (11) | 4 (6) | 14 (24) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (6) | 1 (1) | 8 (10) | 3 (3) | 1 (1) | 3 (4) | 6 (8) | 7 (8) | 11 (13) | 6 (7) | 8 (9) | 9 (11) | 4 (4) | 16 (22) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0) | 4 (7) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (5) | 7 (12) | 2 (2) | 3 (3) | 6 (6) | 0 (0) | 8 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 10 (10) | 5 (5) | 2 (2) | 2 (2) | 7 (8) | 9 (11) | 12 (13) | 7 (7) | 12 (12) | 11 (12) | 7 (8) | 13 (18) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 2 (2) | 5 (5) | 2 (3) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sputum purulent (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 1 (2) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 8 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron binding capacity total decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 6 (6) | 4 (4) | 0 (0) | 7 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 6 (6) | 4 (5) | 3 (3) | 2 (2) | 7 (7) | 2 (2) | 5 (6) | 6 (6) | 10 (12) | 8 (9) | 6 (6) | 11 (12) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 3 (6) | 2 (2) | 5 (7) | 2 (4) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 3 (5) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 3 (4) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 1 (2) | 1 (2) | 1 (1) | 5 (10) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asterixis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 4 (5) | 7 (7) | 7 (7) | 3 (3) | 7 (7) | 3 (4) | 15 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 4 (4) | 4 (5) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Poor quality sleep (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital burning sensation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 1 (2) | 4 (5) | 4 (4) | 5 (5) | 1 (1) | 3 (4) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal ventricle prolapse (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 5 (5) | 4 (4) | 1 (1) | 7 (7) | 3 (3) | 5 (5) | 5 (5) | 4 (4) | 7 (7) | 7 (7) | 4 (4) | 17 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin maceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT04032704/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/04/NCT04032704/SAP_001.pdf